CLINICAL TRIAL: NCT07113938
Title: Assessing the Efficacy and Impact of Ambient AI Scribes in Healthcare: A Randomized Controlled Trial
Brief Title: Assessing the Efficacy and Impact of Ambient AI Scribes in Healthcare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Scott Adams, Assistant Professor, Department of Medical Imaging, University of Saskatchewan, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5336
Record Dates: First submitted 2025-07-21; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Use of Ambient AI Scribes; Patient-Phyisican Interaction; Physician Workload; Physician Burnout
Keywords: artificial intelligence; physician workload; physician burnout; documentation quality

STUDY DESIGN:
Masking Description: Two blinded reviewers will independently review each clinical note and assign a PDQI-9 score according to the nine attributes that measure various aspects of documentation quality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient AI Scribe Users (Experimental): This group will make use of the ambient AI scribe in their clinical visits to generate clinical notes for them over the duration of the study.
  Interventions: Device: Ambient AI Scribe
- Non-Ambient AI Users (No Intervention): This group will continue to generate their own clinical notes without the use of ambient AI scribes over the duration of the study.

INTERVENTIONS:
Device: Ambient AI Scribe — Software that records audio of a clinical interaction and generates a clinical note.
  Arms: Ambient AI Scribe Users

SUMMARY:
The goal of this clinical trial is to assess the impacts of ambient AI scribes on the workload and burnout in physicians who see patients in a clinic setting at least twice in a week, as well as the impacts on patient-physician interaction.

The main questions it aims to answer are:

* What is the impact of ambient AI scribe use on physician workload and burnout?
* What is the impact of ambient AI scribe use on quality of patient-physician interaction?

Researchers will compare the group of physicians using the ambient AI scribes to the group not using ambient AI scribes to see if there are any significant differences.

Participants randomly assigned to Group A will make use of the AI scribe and participants randomly assigned to Group B will not use any AI scribe for the 10 working day duration of the study. They will be asked to complete a survey assessing workload and burnout immediately prior to the commencement of the study and at the end of each week of the study or 5 full working days for part time physicians. They will also invite their patients to complete a survey assessing their experience after each clinical interaction.

ELIGIBILITY:
Inclusion Criteria:

* Physicians from family medicine or any specialty
* Physicians who regularly see patients in a clinic setting at least 2 days per week

Exclusion Criteria:

* Physicians who are planning to leave their practice during the study period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Physician Workload as Measured Using the NASA Task Load Index | From enrolment to the end of the study at 10 working days.
  The NASA-TLX is separated into six 100-point scales with 5-point steps that assess mental demand, physical demand, temporal demand, performance, effort, and frustration. A higher score indicates that they feel a greater degree of each of the domains.
Physician Burnout as Measured Using the MBI - HSS (MP) | From enrolment to the end of the study at 10 working days.
  The MBI-HSS (MP) is created specifically for medical personnel and assesses emotional exhaustion (9 items), depersonalization (5 items), and personal accomplishment (8 items).
Quality of Patient-Physician Interaction As Measured Using the CARE Patient Feedback Measure Domain of "Really Listening" | Throughout study completion at 10 working days.
  The CARE measure consists of a series of 10 questions asked of patients with our focus on the domain of whether the physician was "really listening (paying close attention to what you were saying; not looking at the notes or computer as you were talking)" scored on a 5 point Likert scale.

SECONDARY OUTCOMES:
Documentation Quality as Measured by the PDQI-9 | From enrollment to the completion of the study at 10 working days.
  Documentation is scored by two blinded reviewers on a scale from 1-5 (with 5 indicating a higher quality) across 9 domains: up-to-date, accurate, thorough, useful, organized, comprehensible, succinct, synthesized, and internally consistent.
Time Spent Within the EMR for Each Clinical Note | From enrollment to the completion of the study at 10 working days.
  The amount of time spent within the EMR for each clinical note and the amount of time spent editing the note on the ambient AI platform will be tracked using EMR logs and time-tracking tools.
Time Spent in the EMR After Hours | From enrollment to the completion of the study at 10 working days.
  The amount of time spent using the EMR after regular working hours will be measured using EMR logs and time-tracking tools.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Adams, MD, PhD, MEd, FRCPC, Principal Investigator — University of Saskatchewan College of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li B, Crampton N, Yeates T, Xia Y, Tian X, Truong KN. Automating Clinical Documentation with Digital Scribes: Understanding the Impact on Physicians. In: CHI '21: Proceedings of the 2021 CHI Conference on Human Factors in Computing Systems. Association for Computing Machinery; 2021. Accessed July 1, 2024. https://doi.org/10.1145/3411764.3445172
- [Background] Davenport T, Kalakota R. The potential for artificial intelligence in healthcare. Future Healthc J. 2019 Jun;6(2):94-98. doi: 10.7861/futurehosp.6-2-94. PMID 31363513
- [Background] Saag HS, Shah K, Jones SA, Testa PA, Horwitz LI. Pajama Time: Working After Work in the Electronic Health Record. J Gen Intern Med. 2019 Sep;34(9):1695-1696. doi: 10.1007/s11606-019-05055-x. No abstract available. PMID 31073856
- [Background] Tierney AA, Gayre G, Hoberman B, et al. Ambient Artificial Intelligence Scribes to Alleviate the Burden of Clinical Documentation. NEJM Catal. 2024;5(3). doi:10.1056/cat.23.0404
- [Background] Shanafelt TD, Dyrbye LN, West CP, Sinsky CA. Potential Impact of Burnout on the US Physician Workforce. Mayo Clin Proc. 2016 Nov;91(11):1667-1668. doi: 10.1016/j.mayocp.2016.08.016. No abstract available. PMID 27814840